CLINICAL TRIAL: NCT05070650
Title: Efficacy and Safety of the Combination of Acetylcysteine, Paracetamol and Phenylephrine for the Treatment of Common Cold: a Prospective, Randomized, Double-blind, Controlled Trial
Brief Title: Efficacy and Safety of the Combination of Acetylcysteine, Paracetamol and Phenylephrine for the Treatment of Common Cold
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sandoz has decided to withdraw the clinical study due to internal business reasons. No patients were enrolled in any of the participating countries.
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAN-0657
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Acetylcysteine; Acetaminophen; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetylcysteine/Paracetamol/Phenylephrine 200 mg/500 mg/10 mg granules for oral solution (Experimental): Acetylcysteine/Paracetamol/Phenylephrine 200 mg/500 mg/10 mg granules for oral solution: one sachet three times per day
  Interventions: Drug: Acetylcysteine; Drug: Paracetamol; Drug: Phenylephrine
- Paracetamol/Phenylephrine 500 mg/10 mg granules for oral solution (Active Comparator): Paracetamol/Phenylephrine 500 mg/10 mg granules for oral solution: one sachet three times per day
  Interventions: Drug: Paracetamol; Drug: Phenylephrine

INTERVENTIONS:
Drug: Acetylcysteine — 200 mg/500 mg/10 mg granules for oral solution: one sachet three times per day
  Arms: Acetylcysteine/Paracetamol/Phenylephrine 200 mg/500 mg/10 mg granules for oral solution
Drug: Paracetamol — 500 mg/10 mg granules for oral solution: one sachet three times per day
Drug: Phenylephrine — 500 mg/10 mg granules for oral solution

SUMMARY:
Prospective, randomized, multinational, multicenter, double-blind trial in 2 parallel groups of patients

DETAILED DESCRIPTION:
This study is a prospective, randomized, multinational, multicenter, double-blind trial in 2 parallel groups of patients.

Patients will undergo screening examinations at Visit 1.

Patients who meet all of the inclusion and none of the exclusion criteria will be randomized to double-blind treatment with one of the following:

* Group A: Acetylcysteine/Paracetamol/Phenylephrine: one sachet three times per day OR
* Group B: Paracetamol/Phenylephrine 500 mg/10 mg granules for oral solution: one sachet three times per day.

A control visit (Visit 2) is planned on Day 3 of treatment.

After the end of the double-blind treatment phase, the patients will undergo an end-of-treatment (EOT) examination at Visit 3 on Day 6.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 75 years inclusive on the date of consent
2. No fever or (mild) fever below 38.5° C
3. Total score (sum of all ratings) of 2 or higher based on the rating of the following symptoms of common cold (Jackson scale):

   1. Sneezing
   2. Nasal discharge
   3. Nasal obstruction
   4. Sore throat
   5. Cough
   6. Headache
   7. Malaise
   8. Chilliness according to the following rating scale: 0 = absent, 1 = mild, 2 = moderate, or 3 = severe
4. Presence of cough with thick mucus production
5. Informed consent to participate in the trial provided in written form

Exclusion Criteria:

1. Duration of any of the symptoms of common cold of more than 72 hours at the time of screening
2. History of hypersensitivity or intolerance to the active substances or any of the excipients of the trial medication
3. Known bronchial asthma or chronic obstructive pulmonary disease
4. Known duodenal or gastric ulcer
5. Known hyperthyroidism
6. Known narrow angle glaucoma
7. Known pheochromocytoma
8. Known prostate adenoma with urine retention
9. Known severe liver failure (Child-Pugh > 9)
10. Known severe cardio-vascular diseases
11. Known porphyria
12. Known glucose-6-phosphate dehydrogenase deficiency
13. High fever (body temperature above 38.5°C)
14. Intake of antibiotics, immunosuppressing, immuno-stimulating or immuno-modulating medication, within 30 days prior to screening visit
15. Intranasal or systemic use of corticosteroids within 30 days prior to screening visit
16. Intake of antihistamines or nasal decongestants within 48 hours prior to screening visit
17. Vaccination within 14 days prior to screening visit
18. Immunocompromised state
19. Suspicion for acute bacterial infection
20. Pregnant or breast-feeding female patient
21. Female patient of childbearing potential (not surgically sterilized/ hysterectomized or postmenopausal for at least 1 year) who is not currently using (documented at screening visit) and not willing to use medically reliable methods of contraception for the entire trial duration such as barrier method, oral, injectable or implantable contraceptives, intrauterine contraceptive devices (IUD), sexual abstinence or vasectomized partner
22. Any other condition of the patient (e.g. serious or unstable medical or psychological condition, acute psychosis) that in the opinion of the investigator may compromise evaluation of the trial treatment or may jeopardize patient's safety, compliance or adherence to protocol requirements
23. Participation in ANY research study involving another investigational medicinal product (IMP) within 30 days prior to screening visit, or simultaneous participation in another clinical study or previous participation in present study
24. Suspected alcohol/ drug dependence or abuse (including heavy smoking: ≥ 20 cigarettes daily)
25. Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the trial
26. Subjects who are known or suspected:

    * not to comply with the trial directives
    * not to be reliable or trustworthy
    * to be a dependent person, e.g. a relative, family member, or member/ employee of the investigator's or sponsor's staff
    * subject is in custody or submitted to an institution due to a judicial order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the daily Score of 8 symptoms related to mucus production (SUM8) | Baseline, Day 5
  Score of 8 symptoms related to mucus production (SUM8) will be assessed by the patient in a patient's diary at screening (this will constitute the baseline value) and daily on each day of treatment until and including Day 5. For assessing SUM8 the patients will have to answer questions about their cough and phlegm status. The SUM8 consisted of the sum of the answers to the eight core questions. For calculating the SUM8 the lowest rating corresponds to 0 and highest rating corresponds to 4, with 4 representing the greatest severity of symptoms. The SUM8 thus had a scale range of 0-32 with 0 representing best possible symptoms, and 32 representing greatest severity of symptoms.

SECONDARY OUTCOMES:
Number of adverse events and serious adverse events | Until Day 6, or earlier in case of premature termination
  Assessment of safety and tolerability of the investigational medicinal product against the comparator product for the treatment of common cold
Time to onset of action | Day 1 to Day 5
  Time to onset of action defined as first day of treatment with investigational product on which SUM8 shows statistically significant difference from the comparator product will be reported
Score of 8 symptoms related to mucus production (SUM8) development over the course of the study | Baseline, Day 1 to Day 5
  Score of 8 symptoms related to mucus production (SUM8) will be assessed by the patient in a patient's diary at screening (this will constitute the baseline value) and daily on each day of treatment until and including Day 5. For assessing SUM8 the patients will have to answer questions about their cough and phlegm status. The SUM8 consisted of the sum of the answers to the eight core questions. For calculating the SUM8 the lowest rating corresponds to 0 and highest rating corresponds to 4, with 4 representing the greatest severity of symptoms. The SUM8 thus had a scale range of 0-32 with 0 representing best possible symptoms, and 32 representing greatest severity of symptoms.
Assessment of separate items of Score of 8 symptoms related to mucus production (SUM8) | Baseline, Day 1 to Day 5
  Score of 8 symptoms related to mucus production (SUM8) will be assessed by the patient in a patient's diary at screening (this will constitute the baseline value) and daily on each day of treatment until and including Day 5. For assessing SUM8 the patients will have to answer questions about their cough and phlegm status. The SUM8 consisted of the sum of the answers to the eight core questions. For calculating the SUM8 the lowest rating corresponds to 0 and highest rating corresponds to 4, with 4 representing the greatest severity of symptoms. The SUM8 thus had a scale range of 0-32 with 0 representing best possible symptoms, and 32 representing greatest severity of symptoms.
Sum of changes from baseline in the daily Wisconsin Upper Respiratory Symptom Survey (WURSS-21) | Baseline, Day 1 to Day 5
  The Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) Questionnaire is an evaluative illness-specific outcomes instrument designed to assess the severity of cold symptoms and the impact of the common cold (range 0-140), with higher scores indicating more symptoms and functional impairment.
Assessment of separate items of Wisconsin Upper Respiratory Symptom Survey (WURSS-21) | Baseline, Day 1 to Day 5
  The Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) Questionnaire is an evaluative illness-specific outcomes instrument designed to assess the severity of cold symptoms and the impact of the common cold (range 0-140), with higher scores indicating more symptoms and functional impairment.
Percentage of responders and non-responders to treatment | On Day 3, and after the end of treatment on Day 6
  Percentage of responders and non-responders to treatment based on the assessment of overall response to treatment by the investigator will be reported.

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.